CLINICAL TRIAL: NCT02644759
Title: Efficacy and Safety of Transplantation of Autologous Stem Cells Into Pancreatic Artery, Combined With Immunomodulation for the Treatment of Type 1 Diabetes Mellitus
Brief Title: Transplantation of Autologous Stem Cells for the Treatment of Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stem Cells Arabia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCA-DM1
Record Dates: First submitted 2015-12-21; First posted 2016-01-01 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Diabetes Mellitus Type 1; Autoimmune Diseases; Endocrine System Diseases; Glucose Metabolism Disorders; Immune System Diseases; Metabolic Diseases
Keywords: Stem Cells; Transplantation; Immunomodulation; CD34; CD133; ClinicMACS
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Autoimmune Diseases; Endocrine System Diseases; Glucose Metabolism Disorders; Immune System Diseases; Metabolic Diseases | interventions — Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stem Cell Transplantation (Experimental): Interventional radiology-mediated transplantation of purified, autologous stem cells into pancreatic artery and capillaries, and intravenous injection of autologous, immunomodulated mononuclear cells.
  Interventions: Biological: Stem Cell Transplantation

INTERVENTIONS:
Biological: Stem Cell Transplantation — Interventional radiology-mediated transplantation of purified, autologous stem cells into pancreatic artery and capillaries, and intravenous injection of autologous, immunomodulated mononuclear cells.

SUMMARY:
Type 1 diabetes mellitus (T1DM) is a chronic, autoimmune condition that involves the progressive destruction of pancreatic β-cells, eventually resulting in the loss of insulin production and secretion. Hence, an effective treatment for T1DM should focus on controlling anti-β-cell autoimmunity, combined with regeneration of lost pancreatic β-cell populations, with minimal risk to the patient.

This is a phase I and II clinical trial for treatment of patient with confirmed diagnosis of T1DM for at least 12 months prior to enrolment in this trial. This study aims to determine the combined effects of autologous stem cell transplantation and immunomodulation, on regeneration of lost β-cells and halting the immune attack on the pancreatic β-cells, respectively.

DETAILED DESCRIPTION:
Patients with T1DM depend on administration of exogenous insulin for survival and for control of long-term complications. The best-established treatment is constricted control of blood glucose accomplished by regular daily injections or constant subcutaneous infusion of insulin as intensive insulin therapy. Although insulin therapy has advanced immensely, even the most modern technologies do not allow the maintenance of normal glucose levels.

This is a prospective pilot study intended to treat patients with T1DM after at least one year of confirmed diagnosis. This study encompasses a two-arm approach; the first arm is composed of clinical-grade purification of autologous, leukapheresis-derived, Cluster of differentiation 34+ and 133+ stem cells (accomplished by utilisation of CliniMACS System and approved clinical-grade Microbeads and accessories), and transplantation of the purified ell populations into pancreatic artery and capillaries via interventional radiology techniques; while the second arm aims at halting the immune attack on pancreatic β-cells through immunomodulation, and is composed of incubation of patient's leukapheresis with cord blood-derived mesenchymal stem cells for 3-6 hours, and return of the patient's own white blood cells back into the patient via intravenous injection. Patients are first mobilised with 10 ug/Kg Granulocyte-Colony Stimulating Factor (GCSF) for five day, and then Mononuclear Cells are collected from the patient via leukapheresis.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed Type 1 diabetes mellitus diagnosed for at least 12 months prior to execution of this protocol.

Exclusion Criteria:

* Pregnancy
* Severe psychiatric disorder
* Severe organic impairment (renal, hepatic, cardiac, pulmonary)
* Active infectious disease
* Previous or present neoplastic disease
* Any serious complications due to poor control of diabetes, including: lower limb ischemia, kidney failure, liver failure, vision impairment, peripheral neuropathies, poor circulation.

Ages: 8 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2014-02; Primary Completion 2017-08 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Exogenous insulin dose | 1 month

SECONDARY OUTCOMES:
Anti-GAD titres | 1 month, 3 months, 6 months, 12 months, 24 months, 36 months
C-peptide level | 1 month, 3 months, 6 months, 12 months, 24 months, 36 months
HbA1c level | 1 month, 3 months, 6 months, 12 months, 24 months, 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Stem Cells Arabia, Amman, Jordan